CLINICAL TRIAL: NCT06451601
Title: The Metabolic and Respiratory Effects of Intermittent Hypoxia-hyperoxia Therapy in Obese Patients Within the Complex Management of Medical Rehabilitation
Brief Title: Intermittent Hypoxia-hyperoxia Therapy in Obese Patients (IHHTOP)
Acronym: (IHHTOP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Balnear and Rehabilitation Sanatorium Techirghiol (Other)
Responsible Party: Principal Investigator, Elena-Valentina Ionescu, Assit. Prof. Dr. Ionescu Elena Valentina, Balnear and Rehabilitation Sanatorium Techirghiol
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AndreeaUzun
Record Dates: First submitted 2024-05-24; First posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Obesity
Keywords: intermittent hypoxia hyperoxia therapy; metabolic effects; respiratory effects; medical rehabilitation
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IHHT Group (Experimental): IHHT group with 35 patients: The patients in the IHHT group underwent intermittent hypoxia-hyperoxia therapy using the CellOxy Device.Initially, patients performed hypoxic tests 1 and 2, to determine the optimal oxygen level and to be included in a typology (type I, II, or III).
  Starting from the following day, patients in the IHHT group were subjected to intermittent hypoxia-hyperoxia as follows: hypoxia with 9-16% O2 for 5-7 minutes, followed by exposure to hyperoxia with ~35% O2 for 2-5 minutes.
  In total, patients in the IHHT group performed 9 sessions of hypoxic-hyperoxic therapy: testing on the first day (hypoxic tests 1 and 2), followed by 4 days of sessions in the first week, 2 days of rest on the weekend and then another 5 days of sessions in the second week. Simultaneously with the intermittent hypoxia-hyperoxia therapy, the patients benefited from complex balneo-physical-kinetic treatment.
  Interventions: Device: Intermittent hypoxia-hyperoxia therapy
- Control Group (Active Comparator): Control group with 35 patients: The control group completed only the comprehensive balneo-physical-kinetic treatment (hydrokinetotherapy and hydrothermotherapy using specific natural environmental factors: sapropelic mud and salt water from Lake Techirghiol, electrotherapy, massage therapy and kinetotherapy), without intermittent hypoxia-hyperoxia therapy, neither real nor simulated.
  Interventions: Device: Intermittent hypoxia-hyperoxia therapy

INTERVENTIONS:
Device: Intermittent hypoxia-hyperoxia therapy — Data on demographics and clinical conditions was gathered. The investigators collect the next features: sex, age, occupation, environment, body mass index, nutritional status, abdominal circumference, hip circumference, smoking, alcohol. Also, the patients performed a 6-minute walking test.
  Other Names:
  * Hydrokinetotherapy
  * Hydrothermotherapy
  * Electrotherapy
  * Massage therapy
  * Kinetotherapy

SUMMARY:
Obesity represents the excessive or abnormal accumulation of adipose tissue in the body, which affects health through its association with the risk of developing diabetes mellitus, cardiovascular and pulmonary diseases and hypertension.

Obesity can cause significant respiratory changes, so obese patients present pulmonary complications more frequently than individuals with normal weight.

Intermittent hypoxia (IH) represents the alternation between repeated episodes of hypoxia interspersed with normoxic episodes. Intermittent hypoxia-hyperoxia is the therapy that uses hyperoxic intervals instead of normoxic ones between hypoxic breathing sessions.

This study aimed to evaluate the effectiveness of intermittent hypoxia-hyperoxia therapy among obese patients, focusing on metabolic and respiratory effects. The study aimed to determine if this method could bring benefits in managing or alleviating the complications associated with obesity.

A total of 70 obese patients will be recruited and randomized to either the IHHT group or the control group. The intervention group will receive IHHT while the control group will not receive this therapy.

All patients will be assessed at baseline and after 2 weeks of treatment using a variety of clinical and functional measures. The study's results will be used to determine whether IHHT benefits the patients who follow it.

This study is designed to contribute to the existing body of knowledge on treating obese patients. The results of the study will be of interest to clinicians, researchers, and patients.

DETAILED DESCRIPTION:
The study was a prospective, randomized controlled, unicentric study conducted at the Balneal and Rehabilitation Sanatorium Techirghiol (BRST) in Romania. A total of 70 obese patients (BMI > 30 kg/m2) were enrolled in the study. The patients were randomly assigned to either the IHHT group or the control group.

Patients in the intervention group received intermittent hypoxia-hyperoxia therapy and patients in the control group did not receive this therapy. Simultaneously with the intermittent hypoxia-hyperoxia therapy, the patients benefited from complex balneo-physical-kinetic treatment which included hydrokinetotherapy and hydrothermotherapy using specific natural environmental factors: sapropelic mud and salt water from Lake Techirghiol, electrotherapy, massage therapy and kinetotherapy.

The 35 patients in the IHHT group underwent intermittent hypoxia-hyperoxia therapy using the CellOxy Device. During the hypoxic phases, patients received concentrations of 9-16% O2, while during the hyperoxic phases, approximately 35% O2 was administered.

During both testing and actual therapy sessions, patients remained in a comfortable position, lying on a bed. Initially, patients performed hypoxic tests 1 and 2, to determine the optimal oxygen level and to be included in a typology (type I, II, or III). Based on the obtained data, the device automatically calculated and planned personalized IHHT sessions for each patient.

Starting from the following day, patients in the IHHT group were subjected to intermittent hypoxia-hyperoxia as follows: hypoxia with 9-16% O2 for 5-7 minutes, followed by exposure to hyperoxia with ~35% O2 for 2-5 minutes. During the sessions, both SpO2 and heart rate were constantly monitored using the device's built-in pulse oximeter.

In total, patients in the IHHT group performed 9 sessions of hypoxic-hyperoxic therapy: testing on the first day (hypoxic tests 1 and 2), followed by 4 days of sessions in the first week, 2 days of rest on the weekend and then another 5 days of sessions in the second week.

The initial assessment of patients consisted of a comprehensive medical examination, which identified their comorbidities, family history, verification of medication for associated pathologies and behavioral factors (smoking, alcohol consumption, psychosocial stress).

All patients underwent the following measurements: resting blood pressure (BP), heart rate (HR), blood oxygen saturation (SpO2), anthropometric data: height (cm), body weight (kg), waist circumference (cm), and hip circumference (cm), BMI calculation, blood sampling (urea, uric acid, creatinine, glucose, total cholesterol, AST, ALT). Regardless of the presence or absence of changes in the analysis results, patients were included in the study. We consider it important to investigate the entire spectrum of the studied patients, including those with evident changes in their analyses and those with normal results, to obtain a comprehensive and representative image of the researched phenomenon. The patients also performed a 6-minute walk test and a spirometry.

After completing the 2 weeks of treatment at the Balneal and Rehabilitation Sanatorium of Techirghiol, the final assessment identified the same parameters as followed initially.

The statistical analysis was performed using IBM SPSS statistics software version 25. Data are presented as mean ± standard deviation (SD) for continuous variables in case of symmetric distributions, median and IQR (Interquartile range IQR = P75-P25) for numerical discrete variables or for continuous variables in case of skewed distributions, or as frequencies and percentages for categorical variables. The normality of the continuous data was estimated with Shapiro-Wilk Tests of Normality. For hypotheses testing: Independent Samples Mann Whitney U test, Related Samples Wilcoxon Signed Rank Test, Chi-Square Test of association, were used depending on the type of analyzed variables. Spearman's correlation coefficient was used as a statistical measure of the strength of a relationship between paired data. The significance level α was set at 0.05. If the test statistic for every conducted test was in the critical region, and the p-value was less than or equal to the significance level, we decided to reject the null hypothesis in favor of the alternative hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* patients with BMI >30 kg/m2
* aged between 40-75 years
* patients to sign the informed consent form
* patients to be compensated and to have medical treatment for associated pathologies

Exclusion Criteria:

* BMI <30 kg/m2
* age under 40 or over 75 years
* refusal to sign the informed consent form
* patients presenting contraindications to intermittent hypoxia-hyperoxia therapy
* patients presenting contraindications to complex medical rehabilitation treatment

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-05-06 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
Metabolic effects | Two measurements, at the beginning of treatment and after 2 weeks of treatment.
  Blood sampling (urea, uric acid, creatinine, glucose, total cholesterol). The Units of Measure for these biomarkers = mg/dL.
Metabolic effects | Two measurements, at the beginning of treatment and after 2 weeks of treatment.
  Blood sampling (AST, ALT). The Units of Measure for these biomarkers = U/L.

SECONDARY OUTCOMES:
Respiratory effects | Two measurements, at the beginning of treatment and after 2 weeks of treatment.
  Spirometry (FVC, FEV1). The Units of Measure = l.
Respiratory effects | Two measurements, at the beginning of treatment and after 2 weeks of treatment.
  Spirometry (FEV1/FVC ). The Units of Measure = %.

CONTACTS AND LOCATIONS:
Locations (1):
- Balneal and Rehabilitation Sanatorium Techirghio, Techirghiol, Constanța County, Romania

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Chamarthi VS, Daley SF. Comprehensive Assessment and Diagnosis of Metabolic and Biomechanical Complications in Obesity. 2025 Aug 29. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK459357/ PMID 29083734
- [Background] Lin X, Li H. Obesity: Epidemiology, Pathophysiology, and Therapeutics. Front Endocrinol (Lausanne). 2021 Sep 6;12:706978. doi: 10.3389/fendo.2021.706978. eCollection 2021. PMID 34552557
- [Background] Thompson WG, Cook DA, Clark MM, Bardia A, Levine JA. Treatment of obesity. Mayo Clin Proc. 2007 Jan;82(1):93-101; quiz 101-2. doi: 10.4065/82.1.93. PMID 17285790
- [Background] Bischoff SC, Schweinlin A. Obesity therapy. Clin Nutr ESPEN. 2020 Aug;38:9-18. doi: 10.1016/j.clnesp.2020.04.013. Epub 2020 May 11. PMID 32690184
- [Background] Dixon AE, Peters U. The effect of obesity on lung function. Expert Rev Respir Med. 2018 Sep;12(9):755-767. doi: 10.1080/17476348.2018.1506331. Epub 2018 Aug 14. PMID 30056777
- [Background] Collins LC, Hoberty PD, Walker JF, Fletcher EC, Peiris AN. The effect of body fat distribution on pulmonary function tests. Chest. 1995 May;107(5):1298-302. doi: 10.1378/chest.107.5.1298. PMID 7750322
- [Background] Hegewald MJ. Impact of obesity on pulmonary function: current understanding and knowledge gaps. Curr Opin Pulm Med. 2021 Mar 1;27(2):132-140. doi: 10.1097/MCP.0000000000000754. PMID 33394747
- [Background] Beuther DA, Sutherland ER. Overweight, obesity, and incident asthma: a meta-analysis of prospective epidemiologic studies. Am J Respir Crit Care Med. 2007 Apr 1;175(7):661-6. doi: 10.1164/rccm.200611-1717OC. Epub 2007 Jan 18. PMID 17234901
- [Background] Ford ES, Cunningham TJ, Mercado CI. Lung function and metabolic syndrome: Findings of National Health and Nutrition Examination Survey 2007-2010. J Diabetes. 2014 Nov;6(6):603-13. doi: 10.1111/1753-0407.12136. PMID 26677470
- [Background] Burtscher M, Gatterer H, Szubski C, Pierantozzi E, Faulhaber M. Effects of interval hypoxia on exercise tolerance: special focus on patients with CAD or COPD. Sleep Breath. 2010 Sep;14(3):209-20. doi: 10.1007/s11325-009-0289-8. Epub 2009 Aug 18. PMID 19688232
- [Background] Glazychev OS. [Optimization of clinical application of interval hypoxic training]. Med Tekh. 2013 May-Jun;(3):21-4. No abstract available. Russian. PMID 24003497
- [Background] Uzun AB, Iliescu MG, Stanciu LE, Ionescu EV, Ungur RA, Ciortea VM, Irsay L, Motoasca I, Popescu MN, Popa FL, Pazara L, Tofolean DE. Effectiveness of Intermittent Hypoxia-Hyperoxia Therapy in Different Pathologies with Possible Metabolic Implications. Metabolites. 2023 Jan 25;13(2):181. doi: 10.3390/metabo13020181. PMID 36837800
- [Background] Glazachev OS, Zvenigorodskaia LA, Dudnik EN, Iartseva LA, Mishchenkova TV, Platonenko AV, Spirina GK. [Interval hypoxic-hyperoxic training in the treatment of the metabolic syndrome]. Eksp Klin Gastroenterol. 2010;(7):51-6. Russian. PMID 21033083
- [Background] Costalat G, Lemaitre F, Tobin B, Renshaw G. Intermittent hypoxia revisited: a promising non-pharmaceutical strategy to reduce cardio-metabolic risk factors? Sleep Breath. 2018 Mar;22(1):267-271. doi: 10.1007/s11325-017-1459-8. Epub 2017 Feb 2. PMID 28155101
- [Background] Afina AB, Oleg SG, Alexander AB, Ines D, Alexander Yu S, Nikita VV, Denis ST, Daria GG, Zhang Y, Chavdar SP, Dmitriy VG, Elena AS, Irina VK, Philippe Yu K. The Effects of Intermittent Hypoxic-Hyperoxic Exposures on Lipid Profile and Inflammation in Patients With Metabolic Syndrome. Front Cardiovasc Med. 2021 Aug 27;8:700826. doi: 10.3389/fcvm.2021.700826. eCollection 2021. PMID 34513946
- [Background] https://www.cell-oxy.com/thedevice
- [Background] Cortes-Telles A, Ortiz-Farias DL, Pou-Aguilar YN, Almeida-de-la-Cruz L, Perez-Padilla JR. Clinical impact of obesity on respiratory diseases: A real-life study. Lung India. 2021 Jul-Aug;38(4):321-325. doi: 10.4103/lungindia.lungindia_701_20. PMID 34259169
- [Background] Zammit C, Liddicoat H, Moonsie I, Makker H. Obesity and respiratory diseases. Int J Gen Med. 2010 Oct 20;3:335-43. doi: 10.2147/IJGM.S11926. PMID 21116339
- [Background] Murugan AT, Sharma G. Obesity and respiratory diseases. Chron Respir Dis. 2008;5(4):233-42. doi: 10.1177/1479972308096978. PMID 19029235
- [Background] Serebrovska ZO, Serebrovska TV, Kholin VA, Tumanovska LV, Shysh AM, Pashevin DA, Goncharov SV, Stroy D, Grib ON, Shatylo VB, Bachinskaya NY, Egorov E, Xi L, Dosenko VE. Intermittent Hypoxia-Hyperoxia Training Improves Cognitive Function and Decreases Circulating Biomarkers of Alzheimer's Disease in Patients with Mild Cognitive Impairment: A Pilot Study. Int J Mol Sci. 2019 Oct 30;20(21):5405. doi: 10.3390/ijms20215405. PMID 31671598
- [Background] Mallet R, Burtcher J, Manukhina E, Downy F, Glazachev O, Serebrovskaya T, et al. Hypoxic-hyperoxic conditioning and demen-tia. Diagn Manage Dement. (2020) 47:745-60. 10.1016/B978-0-12-815854-8.00047-1
- [Background] Behrendt T, Bielitzki R, Behrens M, Herold F, Schega L. Effects of Intermittent Hypoxia-Hyperoxia on Performance- and Health-Related Outcomes in Humans: A Systematic Review. Sports Med Open. 2022 May 31;8(1):70. doi: 10.1186/s40798-022-00450-x. PMID 35639211
- [Background] Bayer U, Glazachev OS, Likar R, Burtscher M, Kofler W, Pinter G, Stettner H, Demschar S, Trummer B, Neuwersch S. [Adaptation to intermittent hypoxia-hyperoxia improves cognitive performance and exercise tolerance in elderly]. Adv Gerontol. 2017;30(2):255-261. Russian. PMID 28575566
- [Background] Dudnik E, Zagaynaya E, Glazachev OS, Susta D. Intermittent Hypoxia-Hyperoxia Conditioning Improves Cardiorespiratory Fitness in Older Comorbid Cardiac Outpatients Without Hematological Changes: A Randomized Controlled Trial. High Alt Med Biol. 2018 Dec;19(4):339-343. doi: 10.1089/ham.2018.0014. Epub 2018 Sep 22. PMID 30251879
- [Background] Glazachev O, Kopylov P, Susta D, Dudnik E, Zagaynaya E. Adaptations following an intermittent hypoxia-hyperoxia training in coronary artery disease patients: a controlled study. Clin Cardiol. 2017 Jun;40(6):370-376. doi: 10.1002/clc.22670. Epub 2017 Mar 21. PMID 28323322
- [Background] Serebrovskaya TV, Xi L. Intermittent hypoxia training as non-pharmacologic therapy for cardiovascular diseases: Practical analysis on methods and equipment. Exp Biol Med (Maywood). 2016 Sep;241(15):1708-23. doi: 10.1177/1535370216657614. Epub 2016 Jul 12. PMID 27407098
- [Background] Bestavashvili A, Glazachev O, Ibragimova S, Suvorov A, Bestavasvili A, Ibraimov S, Zhang X, Zhang Y, Pavlov C, Syrkina E, Syrkin A, Kopylov P. Impact of Hypoxia-Hyperoxia Exposures on Cardiometabolic Risk Factors and TMAO Levels in Patients with Metabolic Syndrome. Int J Mol Sci. 2023 Sep 24;24(19):14498. doi: 10.3390/ijms241914498. PMID 37833946
- [Background] Iliescu MG, Stanciu LE, Uzun AB, Cristea AE, Motoasca I, Irsay L, Iliescu DM, Vari T, Ciubean AD, Caraban BM, Ciufu N, Azis O, Ciortea VM. Assessment of Integrative Therapeutic Methods for Improving the Quality of Life and Functioning in Cancer Patients-A Systematic Review. J Clin Med. 2024 Feb 20;13(5):1190. doi: 10.3390/jcm13051190. PMID 38592012
- [Background] Irsay L, Ungur RA, Borda IM, Tica I, Iliescu MG, Ciubean AD, Popa T, Cinteza D, Popa FL, Bondor CI, Ciortea VM. Safety of Electrotherapy Treatment in Patients with Knee Osteoarthritis and Cardiac Diseases. Life (Basel). 2022 Oct 24;12(11):1690. doi: 10.3390/life12111690. PMID 36362845
- [Background] Ungur RA, Ciortea VM, Irsay L, Ciubean AD, Nasui BA, Codea RA, Singurean VE, Groza OB, Cainap S, Martis Petrut GS, Borda C, Borda IM. Can Ultrasound Therapy Be an Environmental-Friendly Alternative to Non-Steroidal Anti-Inflammatory Drugs in Knee Osteoarthritis Treatment? Materials (Basel). 2021 May 21;14(11):2715. doi: 10.3390/ma14112715. PMID 34064094